CLINICAL TRIAL: NCT01396031
Title: Matched-Status Exercise Program in Patients Undergoing Myeloablative Allogeneic Blood and Marrow Transplantation: A Feasibility Study
Brief Title: Feasibility Study of Exercises for Myeloablative Allogeneic Blood and Marrow Transplantation (BMT) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BMTSC0002; IRB-08529 (Other: Stanford University IRB Approval Number); 97821 (Other: Stanford University Alternate IRB Approval Number); BMTSC0002 (Other: OnCore)
Record Dates: First submitted 2011-07-11; First posted 2011-07-18 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Allogenic Disease
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Excercise (Experimental): Cardiovascular exercise Standing Hip Abduction Step-up/Step-down Wall Slide Sit-to-Stand Activity / Exercise Diary 3 times per week x ~1 month
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy — Standard of care
  Other Names: physiotherapy

SUMMARY:
Blood and marrow transplantation (BMT) is commonly used in the treatment of oncologic and hematologic disorders. Patients undergoing Hematopoietic stem cell transplantation (HSCT) are screened for functional status among other criteria to ensure that they are able to endure the rigorous treatment involved during Hematopoietic stem cell transplantation (HSCT). The patient entering the transplant process is possibly already functionally compromised from their disease, prior cancer treatment, and possible other co-morbidities. Additional factors of the transplantation that compromise the independent functional status of the patient include the high dose preparative regimen, pancytopenia, steroid-related side effects, hospitalization, transplantation complications such as infections, pulmonary alterations, acute and chronic Graft-versus-host Disease (GVHD), pain, decreased nutritional input, and other sequelae of transplantation.

Physical Therapy has been utilized in this population primarily as a supportive therapy to prevent and limit the patient's functional decline. Studies have addressed general and aerobic exercise in this population but there is a paucity of research investigating the benefits of a strength-training program, particularly performed in weight-bearing, in attenuating the detrimental effects of the transplantation on functional status.

This is a feasibility study questioning if an exercise program including weight-bearing strengthening exercises and cardiovascular exercise is practical for the patients to carry out as inpatients. The study will also preliminarily determine if this exercise program influences functional outcomes and level of fatigue. Such outcome measures will include 1) FiveTimes Sit-To-Stand Test, 2) Six-Minute Walk Test, 3) stair performance, 4) Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) and Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scales.

The study population will include patients with lymphomas and acute leukemias undergoing matched-related donor allogeneic myeloablative Blood and marrow transplantation (BMT).

ELIGIBILITY:
Inclusion Criteria:

* All diagnoses admitted for a first allogeneic myeloablative Blood and marrow transplantation (BMT)
* Adult subjects greater or equal to 18 year of age. There are no gender or ethnic restrictions
* Karnofsky performance status >= 70%.
* Admitted to E1 Day-7 (+/- 3 days).
* Patients must be informed of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients with musculoskeletal, neurological, cardiovascular, and pulmonary impairments will be excluded. Cardiovascular and pulmonary status will be confirmed prior to transplantation by electrocardiogram, echocardiogram, and pulmonary function tests. Musculoskeletal and screening for neurological impairments will be assessed by Karnovsky score >=70% and by Physical Therapy assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Effect of implementing a matched-status exercise program in patients undergoing allogeneic myeloablative Blood and marrow transplantation (BMT). | 100 days

SECONDARY OUTCOMES:
Effect of exercise program on functional status in patients. | 100 days
Effect of exercise program on quality of life in patients. | 100 days
Effect of exercise program on fatigue in patients. | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lu, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States